CLINICAL TRIAL: NCT05119543
Title: Refractive Error in Chinese Primary and High School Students Before and Amidst COVID-19 in Tianjin
Brief Title: Refractive Error in Chinese Students
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021022
Record Dates: First submitted 2021-11-01; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Myopia
Keywords: COVID-19; Refractive error; China; Myopia
MeSH Terms: conditions — Myopia; COVID-19; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Grade: The changes in myopia rate in 3 years were compared by generalized estimation equation in different grades
  Interventions: Other: outdoor time

INTERVENTIONS:
Other: outdoor time — This cohort study aimed to assess the change of refractive status in Chinese school children under different outdoor time

SUMMARY:
This cohort study aimed to assess the change of refractive status in Chinese school children.

DETAILED DESCRIPTION:
A cohort study was conducted in 96 primary and secondary schools in 16 districts of Tianjin from 2018 to 2020, including about 36452 people totally. The changes in myopia rate in 3 years were compared by a generalized estimation equation. The distribution of average equivalent spherical mirror and different regions and grades was evaluated by linear regression analysis, and the correlation between the equivalent spherical mirror and different gender, nationality, and age was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* no concurrent eye disease
* age from 6 to 18 years old

Exclusion Criteria:

* significant systemic illnesses
* ocular conditions
* congenital corneal diseases
* pterygium, keratoconus
* corneal degeneration or dystrophy
* media opacity, uveitis, glaucoma
* history of ocular surgery
* neurologic diseases
* retinal disease.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This large-scale cohort study was conducted in 36452 schoolchildren on myopia development among schoolchildren in 96 elementary and high schools in 16 districts of Tianjin in China.
Sampling Method: Non-Probability Sample
Enrollment: 36452 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
refractive error | change from baseline at 36 months
  The changes in refractive error were compared by generalized estimation equation.
sex disparity | change from baseline at 36 months
  The changes in refractive error were compared between different sex

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, director, Study Chair — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

REFERENCES:
- [Background] Saw SM, Matsumura S, Hoang QV. Prevention and Management of Myopia and Myopic Pathology. Invest Ophthalmol Vis Sci. 2019 Feb 1;60(2):488-499. doi: 10.1167/iovs.18-25221. PMID 30707221
- [Background] Wang J, Li Y, Musch DC, Wei N, Qi X, Ding G, Li X, Li J, Song L, Zhang Y, Ning Y, Zeng X, Hua N, Li S, Qian X. Progression of Myopia in School-Aged Children After COVID-19 Home Confinement. JAMA Ophthalmol. 2021 Mar 1;139(3):293-300. doi: 10.1001/jamaophthalmol.2020.6239. PMID 33443542
- [Background] Wang W, Zhu L, Zheng S, Ji Y, Xiang Y, Lv B, Xiong L, Li Z, Yi S, Huang H, Zhang L, Liu F, Wan W, Hu K. Survey on the Progression of Myopia in Children and Adolescents in Chongqing During COVID-19 Pandemic. Front Public Health. 2021 Apr 28;9:646770. doi: 10.3389/fpubh.2021.646770. eCollection 2021. PMID 33996724